CLINICAL TRIAL: NCT04308759
Title: Full Scale Randomized Trial of an Innovative Conversational Agent for Smoking Cessation (QuitBot)
Brief Title: An Innovative Conversational Agent (Quitbot) for Smoking Cessation
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RG1006844; NCI-2020-00136 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RG1006844 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA247156 (NIH); 10359 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-03-06; First posted 2020-03-16 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Cigarette Smoking-Related Carcinoma
Keywords: Smoking; smoking cessation; quitting smoking; chatbot
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (QuitBot Experimental) (Experimental): Participants participate in the Quitbot program for 42 days to support quitting smoking. Therapy description withheld to protect the integrity of the study.
  Interventions: Other: Experimental Smoking Cessation Program
- Group II (QuitBot Control) (Active Comparator): Participants participate in the Quitbot program for 42 days to support quitting smoking. Therapy description withheld to protect the integrity of the study.
  Interventions: Other: Control Smoking Cessation Program

INTERVENTIONS:
Other: Experimental Smoking Cessation Program — Participate in Quitbot experimental cessation program
  Other Names: Experimental
  Arms: Group I (QuitBot Experimental)
Other: Control Smoking Cessation Program — Participate in Quitbot control cessation program
  Other Names: Control
  Arms: Group II (QuitBot Control)

SUMMARY:
This phase III trial compares two remote digital smoking cessation programs to see how well they work for quitting smoking.

DETAILED DESCRIPTION:
OUTLINE:

Participants are randomized to 1 of 2 groups. Both groups receive access to a 42-day quit smoking program.

GROUP I: Experimental program, for 42 days to support quitting smoking. After the completion of study, patients are followed up at 3, 6, and 12 months.

GROUP II: Control program, for 42 days to support quitting smoking. After the completion of study, patients are followed up at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Smokes at least one cigarette a day for the past 12 months
* Wants to quit cigarette smoking within the next 30 days (consistent with text messaging intervention trials)
* If concurrently using any other nicotine or tobacco products, wants to quit using them within the next 30 days
* Interested in learning skills to quit smoking
* Willing to be randomly assigned to either intervention
* Resides in United States (US) and will continue to reside in the US for the next 12 months
* Has at least daily access to their own smartphone
* Has text messaging on their smartphone and knows how to download a smartphone application
* Willing and able to read in English, and
* Not using other smoking cessation interventions (This eligibility requirement helps ensure results are due to the treatments we recommend rather than those that participants are doing on their own.)

Exclusion Criteria:

* The reverse of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1647 (Actual)
Dates: Start 2022-07-24 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with 30-day biochemically confirmed cigarette smoking cessation | At 12 months after randomization
  No smoking at all in the past 30 or more days. Complete the biochemical verification procedure that is mailed (Alere saliva-based smoking cessation verification test).

SECONDARY OUTCOMES:
Number of participants with 30-day biochemically confirmed cigarette smoking cessation | At 3 and 6 months after randomization
  No smoking at all in the past 30 or more days. Complete the biochemical verification procedure that is mailed (Alere saliva-based smoking cessation verification test).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan B. Bricker, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bricker JB, Sullivan BM, Mull KE, Lavista-Ferres J, Santiago-Torres M. Efficacy of a conversational chatbot for cigarette smoking cessation: Protocol of the QuitBot full-scale randomized controlled trial. Contemp Clin Trials. 2024 Dec;147:107727. doi: 10.1016/j.cct.2024.107727. Epub 2024 Oct 28. PMID 39490766

DOCUMENTS (1):
  • Informed Consent Form (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT04308759/ICF_000.pdf